CLINICAL TRIAL: NCT01044940
Title: Measurements of Colloid Osmotic Pressure in Interstitial Fluid and Plasma in Healthy and Sick Children
Status: Completed | Type: Observational
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 093137
Record Dates: First submitted 2010-01-07; First posted 2010-01-08 (Estimated); Last update posted 2015-09-10 (Estimated); Status verified 2015-09

CONDITIONS: Colloid Osmotic Pressure
Keywords: Colloid Osmotic pressure in interstitial fluid; Colloid Osmotic pressure in plasma; Protein fractions in interstitial fluid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and interstitial fluid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Birth asphyxia: Babies suffering from birth asphyxia
- Blood transfusion: Babies who receives blood transfusion
- Heart Surgery: Babies who need heart surgery

SUMMARY:
The purpose of this study is to measure colloid osmotic pressure in interstitial fluid and plasma in healthy children under two years, in asphyxiated babies and in children undergoing heart surgery.

ELIGIBILITY:
Inclusion Criteria:

* Newborn

Exclusion Criteria:

* Syndromes

Ages: 1 Hour to 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Asphyxiated babyes Children with heart defects who need surgery Newborn who need blood transfusion
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2010-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Colloid osmotic pressure | 6, 12, 24, 48, 72 hours post partum

CONTACTS AND LOCATIONS:
Overall Officials: Hans Joergen T Guthe, MD, Principal Investigator — Haukeland University Hospital
Locations (1):
- Haukeland University hospital, Bergen, Bergen, Norway

REFERENCES:
- [Derived] Guthe HJT, Nedrebo T, Damas JK, Wiig H, Berg A. Transcapillary fluid flux and inflammatory response during neonatal therapeutic hypothermia: an open, longitudinal, observational study. BMC Pediatr. 2018 Feb 23;18(1):82. doi: 10.1186/s12887-018-1020-3. PMID 29471782